CLINICAL TRIAL: NCT01436552
Title: Psychopathological Risk Factors Associated With Conversion From Mild Cognitive Impairment to Dementia
Acronym: FPRMCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Jean Pierre Clement, Professor of Psychiatry -Ph.D, Centre Hospitalier Esquirol
Other Study IDs: B1001104-10
Record Dates: First submitted 2011-09-16; First posted 2011-09-19 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2010-02

CONDITIONS: Mild Cognitive Impairment
Keywords: MCI; Depression; Alzheimer; Life events
MeSH Terms: conditions — Cognitive Dysfunction; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background: Dementias (Alzheimer's disease and related syndromes), in their sporadic form, have multifactorial origin. Several risk factors (RF) are currently recognized like the cardiovascular RF, some genes of susceptibility, but the impact [1] of traumatic life events (TLE), considered as psychosocial RF (Persson & Skoog, 1996; Charles et al, 2006), [2] of anxiety and/or depression, [3] of the premorbid personality (Clément et al, 2003) with his coping strategies, and [4] of the lifestyle (which results from the personality), for the moment are still underestimated. Dementia disease can be clinically preceded by a mild cognitive impairment (MCI) (Petersen et al, 1996) which is however potentially reversible.

Purpose: Actually, there is no study concerning the rate of conversion from MCI to dementia according to the presence or not of TLE. The aim of this study is to assess association between TLE and conversion rate from MCI to dementia.

Methods: Patients with MCI will be recruited in different memory clinics (Limoges and others) Primary outcome: Occurrence of dementia according to DSM-IV-TR criteria in MCI patients according to their cumulated score of TLE measured by EVVIE.

Secondary outcomes: Occurrence of dementia in MCI patients according to various other psychopathological factors: anxiety, depression, apathy, personality features, alexithymia and resilience levels and life style.

Study design: Epidemiologic cohort longitudinal and prospective multicenter study.

DETAILED DESCRIPTION:
Eligibility criteria:

* Inclusion criteria:

  * Man or woman ≥ 50 years.
  * Patient with MCI, of any type, according to the criteria of Petersen et al, 2001.
  * Clinical Dementia Rating (CDR) ≤ 0,5.
  * Instrumental activities of daily living (IADL)=0.
  * MMSE > 26.
  * Cognitive and functional capacities well enough in order to avoid a possible diagnosis of Alzheimer's disease based on clinical evidences (DSM-IV TR) cannot be done during initial visit.
  * Ambulatory patient.
  * Visual and auditory capabilities (equipment allowed) and oral or written capacity able for the development of suitable tests (according to the clinician).
* exclusion criteria:

  * Patient with identified neurological problems.
  * Patient with developing and/ or non-stabilized psychiatric disease.
  * Patient with biological disorders observed during diagnostic process. Number of subjects: 392 subjects Statistical analysis: Statistical analyses will be performed by the Unité Fonctionnelle de Recherche Clinique et de Biostatistique from the Limoges teaching hospital using SAS® V 9.1.3 software (SAS Institute Cary, NC). Level of significance will be 0.05 for all analyses. Statistical analyses will be performed and presented in agreement with STROBE guidelines.

Descriptive analyses

Quantitative variables will be described using mean ± standard deviation or median and interquartile range. Qualitative variables will be described using frequencies, percentages and 95% confidence intervals assessed with exact method.

A flow chart of patients will be presented.

Main analysis Association between dementia and EVVIE score will be assessed through relative risk calculation. 95% confidence interval will also be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman ≥ 50 years.
* Patient with MCI, of any type, according to the criteria of Petersen et al, 2001.
* Clinical Dementia Rating (CDR) ≤ 0,5.
* Instrumental activities of daily living (IADL)=0.
* MMSE > 26.
* Cognitive and functional capacities well enough in order to avoid a possible diagnosis of Alzheimer's disease based on clinical evidences (DSM-IV TR) cannot be done during initial visit.
* Ambulatory patient.
* Visual and auditory capabilities (equipment allowed) and oral or written capacity able for the development of suitable tests (according to the clinician).

Exclusion Criteria:

* Patient with identified neurological problems.
* Patient with developing and/ or non-stabilized psychiatric disease.
* Patient with biological disorders observed during diagnostic process.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MCI will be recruited in different memory clinics (Limoges and others)
Sampling Method: Probability Sample
Enrollment: 392 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dementia according to DSM-IV-TR criteria in MCI patients according to their cumulated score of TLE measured by EVVIE. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Clement, MD, PhD, Principal Investigator — CH Esquirol
Locations (1):
- CH Esquirol, Limoges, France